CLINICAL TRIAL: NCT01836146
Title: International First-in-Human Study of the EnligHTN Generation 2 System in Patients With Drug-resistant Uncontrolled Hypertension
Acronym: EnligHTN III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1202
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Artery Ablation (Experimental)
  Interventions: Device: EnligHTN™ Renal Artery Ablation Catheter

INTERVENTIONS:
Device: EnligHTN™ Renal Artery Ablation Catheter

SUMMARY:
The purpose of this First-in-Human Clinical investigation is to evaluate the safety and performance of the St. Jude Medical EnligHTN™ Generation 2 Renal Denervation System for the treatment of patients with drug-resistant uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 and ≤ 80 years of age at time of consent
* Subject must be able and willing to provide written informed consent
* Subject must be able and willing to comply with the required follow-up schedule
* Subject has office Systolic Blood Pressure ≥ 160 mmHg at confirmatory visit
* Subject has a daytime mean Systolic Ambulatory Blood Pressure > 135 mmHg during the two week screening period
* Subject has an office Systolic Blood Pressure that remains ≥160 mmHg despite the stable use of ≥3 antihypertensive medications concurrently at maximally tolerated doses, of which one is a diuretic or subject was previously on diuretic but documented to be diuretic intolerant, for a minimum of 14 days prior to the procedure and with an expectation to maintain for a minimum of 180 days post procedure.

Exclusion Criteria:

* Subject has significant renovascular abnormalities such as renal artery stenosis > 30% in either renal artery
* Subject has undergone prior renal angioplasty, renal denervation, indwelling renal stents, and/or abdominal aortic stent grafts
* Subject has hemodynamically significant valvular heart disease as determined by the Study Investigator
* Subject has a life expectancy less than 12 months, as determined by a Study Investigator
* Subject is participating in another clinical study which has the potential to impact their hypertension management (pharmaceutical/device/homeopathic)
* Subject is pregnant, nursing, or of childbearing potential and is not using adequate contraceptive methods
* Subject has active systemic infection
* Subject has renal arteries with diameter(s) < 4 mm in diameter or <20 mm in length
* Subject has an estimated Glomerular Filtrate Rate (eGFR) <45 mL/min per 1.73 m2 using the Modified Diet in Renal Disease (MDRD) formula
* Subject has Diabetes Mellitus Type I
* Subject has multiple main renal arteries in either kidney
* Subject has an identified secondary cause of hypertension (for example, including, but not limited to, Polycystic kidney disease, Cushing's syndrome, Aldosteronism)
* Subject has evidence of significant abdominal aortic aneurysm (defined as maximum diameter of >4 cm)
* Subject has had a myocardial infarction, unstable angina pectoris or cerebrovascular accident less than 180 days prior to enrollment
* Subject is expected to have cardiovascular intervention within the next 180 days
* Subject has a condition which would interfere with the accurate interpretation of the study objectives including but not limited to a large arm diameter that is unable to accommodate the blood pressure cuff or arrhythmia that interferes with automatic pulse sensing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety Objective | 6 months
  To characterize the rate of serious procedural and device related adverse events from date of procedure through 6 months post procedure, as adjudicated by the Clinical Events Committee (CEC).
Performance objective | 6 months
  To characterize the reduction of office Systolic Blood Pressure at 6 months post procedure as compared to baseline.

SECONDARY OUTCOMES:
Change in Ambulatory Blood Pressure | 1 month, 3 month, 6 month, 12 month, 18 month, 2 years
  Characterization of the change in Ambulatory Blood Pressure parameters over time as compared to baseline
New renal artery stenosis or aneurysm at the site of ablation | 1 month, 3 month, 6 month, 12 month, 18 month, 2 years
  Characterization of renovascular safety as measured by new renal artery stenosis or aneurysm at the site of ablation over time as compared to baseline
Renal Function Change | 1 month, 3 month, 6 month, 12 month, 18 month, 2 years
  Characterization of renal function change over time as compared to baseline as measured by changes in: eGFR, serum creatinine and cystatin C

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (4):
  - St Andrews Hospital, Adelaide, South Australia
  - St. Vincent's Hospital Melbourne, Fizroy, Victoria
  - Monash Heart/Southern Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin